CLINICAL TRIAL: NCT05350826
Title: Targeted Therapies in Chronic Lymphocytic Leukemia and Medico-economic Evaluation of the Ambulatory Medical Assistance Nurse Program : a Prospective Multicenter Randomized Study
Brief Title: Evaluation of the Ambulatory Medical Assistance Nurse Program in Chronic Lymphocytic Leukemia
Acronym: THEMIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/21/0340
Record Dates: First submitted 2022-04-07; First posted 2022-04-28 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Chronic Lymphoid Leukemia
Keywords: Targeted therapy; Ambulatory medical assistance; Chronic lymphoid leukemia; Real-world costs
MeSH Terms: conditions — Leukemia, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambulatory medical assistance (Experimental): Patient benefiting from the ambulatory medical assistance nurse program in addition to conventional care for patients chronic lymphoid leukemia under targeted therapy
  Interventions: Other: Ambulatory medical assistance
- Conventional care (No Intervention): Patient benefiting from conventional care for patients chronic lymphoid leukemia under targeted therapy

INTERVENTIONS:
Other: Ambulatory medical assistance — Ambulatory medical assistance is a patient-empowerment program and consists to programmed phone calls (bi-monthly for the first 6 months then monthly for the following 6 months) delivered by an oncology nurse, in link with the hematologist.
  Arms: Ambulatory medical assistance

SUMMARY:
The emergence of targeted therapy (ibrutinib, venetoclax, acalabrutinib) has revolutionized the management practices of chronic lymphoid leukemia due to their effectiveness. However, targeted therapy induces a significant additional cost compared to treatment with immunochemotherapy and their use can be problematic due to the frequent occurrence of side effects, which can be serious. In order to improve the current management of patients treated with targeted therapy, the aim of this study is to evaluate the ambulatory medical assistance nurse program. Ambulatory medical assistance is based on regular telephone calls to patient's homes by a specialist nurse and consists of the monitoring, detection and early management of possible adverse effects of targeted therapy, in link with the hematologist. The main objective of this clinical research is to determine efficiency of the ambulatory medical assistance nurse program.

DETAILED DESCRIPTION:
This research is a prospective randomized multicenter comparative study in 2 parallel groups (1: 1) : patients benefiting from the ambulatory medical assistance nurse program in addition to conventional care versus patients benefiting from conventional care. For each patient, data will be collected during 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over the age of 18
* Patients with chronic lymphoid leukemia and starting treatment with targeted therapy: ibrutinib, venetoclax or acalabrutinib, alone or in combination with obinutuzumab or rituximab in 1L or R/R according to the indications of the Marketing Authorization.
* Be able to understand the objective and the constraints related to the research
* Patient having signed the consent form
* Patient with Social Security affiliation or equivalent
* Person able to speak on the phone

Exclusion Criteria:

* Patient who has already benefited from ambulatory medical assistance nurse program with a previous treatment
* Pregnant women
* Patients under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Ambulatory medical assistance efficiency | 1 year
  To evaluate at 1 year the efficiency of the ambulatory medical assistance program, through the scale EQ-5D-5L

SECONDARY OUTCOMES:
Survival of patients | 1 and 2 years after initiation of targeted therapy
  Compare the survival of patients with or without ambulatory medical assistance at 1 and 2 years
Quality of life of patients | at inclusion, 1 and 2 years after initiation of targeted therapy
  Compare the quality of life of patients with or without ambulatory medical assistance with European Organisation for Research and Treatment of Cancer C30 scores
Cost-effectiveness analysis | at 1 and 2 years
  Perform a cost-effectiveness analysis at 1 and 2 years comparing costs and survival from a community perspective

CONTACTS AND LOCATIONS:
Overall Officials: Loïc YSEBAERT, MD, PhD, Study Director — University Hospital, Toulouse
Locations (16):
- France (16):
  - CH Sud Réunion, Saint-Pierre, ILE de LA Reunion
  - CHU d'Angers, Angers
  - CHU DE BREST Hôpital A.Morvan, Brest
  - Hôpital Estaing, Clermont-Ferrand
  - CHRU Dijon, Dijon
  - CH du Mans, Le Mans
  - Centre Hospitalier Lyon sud, Lyon
  - Centre Léon Bérard, Lyon
  - Hôpital Emile MULLER, Mulhouse
  - CHRU de Nancy, Nancy
  - Institut de Cancérologie du Gard, Nîmes
  - Hôpital Saint-Louis, Paris
  - CHU de Reims- Hôpital R.Debré, Reims
  - CHU de RENNES, Rennes
  - Hôpital Bretonneau, Tours
  - CH Bretagne Atlantique Vannes, Vannes

IPD SHARING:
Plan to Share IPD: No